CLINICAL TRIAL: NCT02811094
Title: LUMIER² Study : LUpus Molecular Immunomonitoring to Evaluate the Risk of Relapse
Acronym: LUMIER²
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID situation
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-26; 2015-A00981-48 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adult patients with Systemic LupusErythematosus (SLE) (Other): Adult patients with SLE, clinically quiescent and with no change in treatment in the past 3 months, will be included and followed-up for 12 months. Blood samples will be drawn every 3 months during 12 months in the absence of flare. Patients presenting a flare will be sampled at the time of the flare and 1 month later.
  Interventions: Other: polymerase chain reaction (PCR) technique of blood transcriptome analysis

INTERVENTIONS:
Other: polymerase chain reaction (PCR) technique of blood transcriptome analysis — this study (LUMIER2 study) is to test the hypothesis that a test score or prognostic transcriptomic allows to discriminate clinically quiescent or patients who will not present a push of Systemic Lupus Erythematosus

SUMMARY:
We aim to determine the accuracy or blood transcriptomic signatures to predict the occurrence of flares in patients with SLE that are clinically quiescent at inclusion Systemic Lupus Erythematosus (SLE) is a chronic auto-immune disease evolving by flares, with possible organ damage, and periods of remission. Current biological markers of disease activity are not sufficient to predict the occurrence of flares, monitor response to treatment or adapt therapeutic strategies. A previous study on genome-wide whole blood transcriptomic signatures in SLE (Chiche et al, Arthritis Rheumatology 2014) has identified gene panels associated with SLE disease activity

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic auto-immune disease evolving by flares, with possible organ damage, and periods of remission. Current biological markers of disease activity are not sufficient to predict the occurrence of flares, monitor response to treatment or adapt therapeutic strategies. A previous study on genome-wide whole blood transcriptomic signatures in SLE (Chiche et al, Arthritis Rheumatology 2014) has identified gene panels associated with SLE disease activity.

We aim to determine the accuracy or blood transcriptomic signatures to predict the occurrence of flares in patients with SLE that are clinically quiescent at inclusion.

LUMIER² is a prospective multicentric observational study conducted in the departments of Clinical Nephrology, Internal Medicine and Rheumatology in the South of France. Adult patients with SLE, clinically quiescent and with no change in treatment in the past 3 months, will be included and followed-up for 12 months. Blood samples will be drawn every 3 months during 12 months in the absence of flare. Patients presenting a flare will be sampled at the time of the flare and 1 month later.

The inclusion of 300 patients is expected, with a test cohort (150 patients) and a validation cohort (150 patients).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* SLE defined by ACR criteria
* Clinically quiescent disease (SLEDAI =< 4 without clinical flare) and absence of treatment increase in the past 3 months
* Written informed consent

Exclusion Criteria:

* Pregnancy, lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of the blood transcriptomic score to predict SLE flares. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la conception Assistance Publique Hôpitaux de Marseille, Marseille, France